CLINICAL TRIAL: NCT00328887
Title: Phase I, Initial Safety/Toxicity Study on the Transfer of Adenovirus With the CD40 Ligand Gene (AdCUCD40L) to Patients With Stage III or IV Esophageal Carcinoma
Brief Title: Safety Study on the Transfer of the CD40 Ligand Gene (AdcuCD40L) to Patients With Esophageal Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding was obtained for this study. No subject were receruited.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0011004683; 5 R01 CA10198-02 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — CD40 Ligand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD40 Gene Transfer (Experimental): Recruitment will be random from the referral base of the investigators from the popula¬tion of individuals with esophageal cancer defined by the protocol inclu¬sion/exclusion criteria.
  Interventions: Genetic: CD40 Gene Transfer

INTERVENTIONS:
Genetic: CD40 Gene Transfer — gene transfer, intratumoral administration
  Other Names: CD40 Ligand Gene (AdcuCD40L)

SUMMARY:
This a pilot clinical study focused on enhancing the patient's anti-tumor immune response in individuals with esophageal cancer by altering the genetic repertoire of the tumors to express CD40L, an activator of dendritic cells. This will be accomplished by endoscopic administration to the tumors of AdcuCD40L, an adenovirus gene transfer vector expressing the coding sequence of the human CD40L cDNA. This study is designed to assess the hypothesis that it is safe to administer the AdcuCD40L vector to individuals with esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is a deadly disease, with only slow advances in therapy over several decades, despite a rapid increase in incidence. Esophageal cancer is estimated to be the seventh most common malignancy worldwide, with incidence rates reaching epidemic proportions in select regions in Asia and Africa. In the United States, it is estimated that 12,300 new cases were diagnosed in 2000, however, the incidence of adenocarcinoma of the esophagus is currently rising faster than that of any other human malignant tumor in this country. Despite advances in surgical technique, chemotherapy, radiotherapy and early detection, only 12% of patients diagnosed with esophageal cancer will survive more than five years, a cure rate more dismal than that seen with cancers of the breast, prostate, colon, and even lung. Survival following treatment for esophageal cancer is stage dependent. This study is directed towards augmenting host anti-tumor immunity by using gene transfer to activate dendritic cells (DC; cells of our immune system that play a central role in initiating immune responses) in tumors of patients with esophageal cancer. Based on extensive pre-clinical data, two proposed clinical trial protocols will evaluate the concept that transient modification of the genetic repertoire of esophageal tumors to express CD40 Ligand (CD40L; a potent activator of DC) will induce the accumulation of activated DC within the tumor, and the in vivo interaction of DC with the tumor cells/tumor antigens will induce tumor-specific immunity. To assess this concept, an adenovirus (Ad) vector (AdcuCD40L) will be used to transfer and transiently express the human CD40L cDNA in esophageal carcinoma by direct injection into the tumor. Phase I represents a dose escalation study to determine the maximum tolerated dose of the vector and will include 12 individuals with unresectable, stage III or IV esophageal cancer. Phase II is a randomized, double-blinded assessment of biologic efficacy and will include 24 individuals with resectable, stage I-III disease who will be undergoing potentially curative resection. Together, both protocols are designed to assess two hypotheses. First, that it is safe to administer the AdcuCD40L vector to individuals with esophageal cancer. Second, that intratumoral administration of the AdCUCD40L vector will induce both the accumulation, in the tumor and in regional lymph nodes, of activated DC, and CD8+ T cells (and other inflammatory cells), including T cells exhibiting tumor-specific responses, as well as systemic antitumor immunity.

ELIGIBILITY:
Inclusion Criteria:

* Must be capable of providing informed consent
* Males and females, age 18 to 75 years
* Hematocrit > 30%
* WBC < 10,000
* Normal prothrombin, partial thromboplastin time; platelet count > 100,000
* Normal liver-related serum parameters
* Blood urea nitrogen < 60 mg/dL, creatinine < 2.5 mg/dl
* No evidence of active infection of any type, including with adenovirus, hepatitis virus (A, B or C) or human immunodeficiency virus
* No evidence of central nervous system, major psychiatric, musculoskeletal or immune disorder
* No allergy to the vehicle used to suspend the virus or contrast materials used in radiographic procedures
* Fertile or infertile individuals; it will be recommended that fertile individuals utilize barrier birth control measures to prevent pregnancy during and for 1 month following the administration of the vector
* Biopsy proven esophageal cancer; stage IIIB or IV; no chemotherapy for 4 weeks prior to vector dosing; and no chemotherapy or radiation for 4 weeks after vector dosing. Patients must have viable tumor in the esophagus (or gastroesophageal junction). In addition, patients must be (1) be untreated; or, (2) show endoscopic evidence of persistence of disease after treatment with conventional chemotherapy, radiotherapy, or both
* Individuals not receiving experimental medications or participating in another experimental protocol for at least 4 weeks prior to entry to the study.
* The study individual must be able to undergo the procedures in the protocol
* Willingness to participate in the study

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria will be unable to participate in the protocol
* Individuals in whom participation in the study would compromise the normal care and expected progression of their disease
* Individuals receiving corticosteroids or other immunosuppressive medications; previous splenectomy or radiation to the spleen; autoimmune disease
* Recent (less than 6 wk) cerebral vascular accident
* Recent (less than 6 wk) transmural myocardial infarction
* Evidence of infection defined by elevated white blood cell count, temperature > 38.5oC or infiltrate on chest x-ray
* Cervical esophageal cancer
* Gastric cancer (tumor more than 50% in the stomach as determined by endoscopy)
* Lack of viable esophageal tumor (applies only to pretreated patients)
* Pathology other than squamous cell or adenocarcinoma
* Malignant ventricular arrhythmia
* Pregnancy
* Immunodeficiency disease, including evidence of HIV infection
* Current alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Since this is a dose escalation, phase I design to evaluate toxicity, the analysis for this section will be purely descriptive. Adverse events will be considered on an individual basis. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - The Valley Hospital, Ridgewood, New Jersey
  - Weill Medical College of Cornell University, New York, New York

IPD SHARING:
Plan to Share IPD: No